CLINICAL TRIAL: NCT03492697
Title: A Phase 1, Open-label Study In Healthy Subjects To Evaluate The Pharmacokinetics Of Pf-06882961 Following Single Oral Administration Of Immediate Release Tablets And An Immediate Release Oral Solution In The Fed State, And Controlled Release Tablets In The Fed And Fasted States
Brief Title: A Single Dose Crossover Study In Healthy Subjects To Evaluate Different Formulations Of PF-06882961
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C3421003
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — danuglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06882961 (Experimental)
  Interventions: Drug: PF-06882961 Immediate Release Tablet; Drug: PF-06882961 Controlled Release Tablet (long); Drug: PF-06882961 Controlled Release Tablet (short); Drug: PF-06882961 Immediate Release Solution

INTERVENTIONS:
Drug: PF-06882961 Immediate Release Tablet — Immediate Release Tablet
Drug: PF-06882961 Controlled Release Tablet (long) — Controlled Release tablet (long)
Drug: PF-06882961 Controlled Release Tablet (short) — Controlled Release tablet (short)
Drug: PF-06882961 Immediate Release Solution — PF-06882961 Immediate Release solution

SUMMARY:
This open label study will evaluate the pharmacokinetics (PK) following single oral doses of different formulations of PF-06882961, including controlled release (CR) tablets at 2 release rates (long and short duration), an immediate release (IR) oral solution, and IR tablets, in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of nonchildbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive
* Body mass index (BMI) within 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal (including pancreatitis), cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug test.
* History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects within 6 months before screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Subjects who have previously participated in prior studies with PF 06882961 as the investigational product.
* Screening supine BP>=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Screening supine 12 lead ECG demonstrating a QTc interval >450 msec or a QRS interval >120 msec.
* Aspartate aminotransferase (AST) level >= 1.25 × upper limit of normal (ULN);
* Alanine aminotransferase (ALT) level >= 1.25 × ULN;
* Total bilirubin level >=1.5 × ULN;
* TSH > ULN;
* HbA1c >=6.5%.
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in the protocol for at least 28 days after the last dose of investigational product.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2), or subjects with suspected MTC per the investigator's judgement.
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of the protocol.
* Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06882961 | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose in each period
Time to Maximum Observed Plasma Concentration (Tmax) for PF-06882961 | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose in each period
Area under the curve from time zero to last quantifiable concentration for PF-06882961 (AUClast) | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose in each period
Area under the curve from time zero to extrapolated infinite time for PF-06882961 (AUCinf), as data permit | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose in each period
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Observed Plasma Concentration for PF-06882961 at 24 hours post-dose (C24) | 24 hours post dose in each period
Plasma Decay Half-Life (t1/2) for PF-06882961, as data permit | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose in each period
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent clearance (CL/F) for PF-06882961, as data permit | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose in each period
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Calculated as Dose/AUCinf
Peak-to-trough (PTR) ratio for PF-06882961 | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose in each period
  Calculated as ratio of Cmax to C24

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (AEs) | Baseline to at least 28 days after last dose
  Assessment by adverse event monitoring, 12 lead ECGs, vital signs and clinical safety laboratory measurements.
AUClast for PF-06882961 for CR tablet (long) and IR tablet in fed state | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose
AUCinf for PF-06882961 for CR tablet (long) and IR tablet in fed state, as data permit | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose
Cmax for PF-06882961 for CR tablet (long) and IR tablet in fed state | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose
AUClast for PF-06882961 for CR tablet (long) in fed and fasted states | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose
AUCinf for PF-06882961 for CR tablet (long) in fed and fasted states, as data permit | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose
Cmax for PF-06882961 for CR tablet (long) in fed and fasted states | 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 28, 32, 36 and 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3421003&StudyName=A+Phase+1%2C+Open-label+Study+In+Healthy+Subjects+To+Evaluate+The+Pharmacokinetics+Of+Pf-06882961+Following+Single+Oral+Administration+Of+Immediate+Release+Tablets+And+An+Immediate+Release+Oral+Solution+In+The+Fed+State%2C+And+Controlled+Release+Tablets+In+The+Fed+And+Fasted+States